CLINICAL TRIAL: NCT02068417
Title: A Prospective, Randomised, Blinded, Placebo-controlled Pilot Study of the Treatment of Erectile Dysfunction With Extracorporeal Shockwave Therapy (ESWT)
Brief Title: Pilot Study of the Treatment of Erectile Dysfunction (ED) With Extracorporeal Shockwave Therapy (ESWT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It has been decided to improve the inclusion criteria for better study outcome
Sponsor: Storz Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU10/002
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Erectile Dysfunction
Keywords: IIEF score; ED
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shock wave treatment (Active Comparator): Shock waves are applied extracorporeally with 0.1 millijoule per square millimeter (mJ/mm2)
  Interventions: Device: shock waves
- Placebo Shock wave treatment (Placebo Comparator): Shock waves are prohibited to enter the body by placebo stand-off.
  Interventions: Device: shock waves

INTERVENTIONS:
Device: shock waves — extracorporeal shock waves: Verum: 0.1 mJ/mm2 Placebo: placebo stand-off
  Other Names: ESWT; extracorporeal shock wave therapy

SUMMARY:
The objective of the pilot study is to assess the feasibility of a full randomised, placebo-controlled clinical trial.The aim is to demonstrate that penile shockwave application in patients with erectile dysfunction of vascular origin leads to a greater increase in potency than in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction for more than 6 months
* Informed consent
* Positive effect of phosphodiesterase type 5 inhibitor (PDE5i)
* IIEF-15 score less than 20
* No neurological disease
* Stable partnership for more than 3 months
* Age 18-75

Exclusion Criteria:

* Total prostatectomy
* Another reason for ED except for vascular disorder
* Clinically significant hematological disease
* Heart stroke, Arrythmia during the last 6 months
* Cancer during the last 5 years
* Intake of antiandrogen
* ED treatment with the last 7 days
* IIEF score higher than, equal to 20
* Previous shockwave treatment

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Effects of erection problems on the sex life (International Index of Erectile Function (IIEF) Questionnaire) | up to 6 months post treatment

SECONDARY OUTCOMES:
Quality of erection (Quality of Erection Questionnaire) | At screening, 1, 3 and 6 months post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Bethanien Krankenhaus Chemnitz gemeinnützige GmbH, Chemnitz, Germany